CLINICAL TRIAL: NCT04179344
Title: The Usability Testing of the IeHS (Integrated E-healthcare Services) Web-based Application in the Therapy Management of HIV and Tuberculosis in Indonesia: a Concurrent Nested Study Design
Brief Title: Usability Study of IeHS in Indonesia
Status: Completed | Type: Observational
Sponsor: Bekasi City Public Hospital (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Principal Investigator, Lusiana Rusdi Idrus, Pharmacist, Bekasi City Public Hospital
Other Study IDs: IeHS_Indonesia
Record Dates: First submitted 2019-08-01; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Human Immunodeficiency Virus; Tuberculosis; Interpersonal Relations; Mobile Phone Use; Adult
Keywords: Pharmaceutical care; HIV; TB; Internet; Surveys and questionnaires; Humans; Pharmacovigilance
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis; Cell Phone Use

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Integrated e-healthcare services (IeHS) web-based app: This usability study is conducted under 3 steps: IeHS simulation, user experience survey using SUS questionnaire, and qualitative study through the in-depth interview.
  Interventions: Other: Integrated e-healthcare services (IeHS) web-based app

INTERVENTIONS:
Other: Integrated e-healthcare services (IeHS) web-based app — Each participant is asked to complete study tasks using the IeHS web-based app as a part of IeHS simulation. This activity is followed by user experience survey, and an in-depth interview to explore user satisfaction on the IeHS web-based app

SUMMARY:
Technology that has a particular focus on patients' needs and ease-of-use and -access plays a significant role in the development of e-health and m-health. The proposed model of a secured mobile health application may promote patient's self-management and enhances adherence in chronic therapy exactly as it is easy-to-use, reducing patient's burden in accessing medication information and instructions, and providing the opportunity for direct communications with health providers in charge for each patient with access to mobile technologies. Consequently, medication errors and unnecessary paperwork in the healthcare system will be avoided as well as giving more time for healthcare providers to pay greater attention to delivering medical care effectively and efficiently.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the world's leading infectious threat as it kills more than 1 million people worldwide every year, with most of them in low and middle-income countries1. Several medical conditions impair innate and acquired immunity and favor the occurrence of TB disease in individuals who are latently infected2,3. People living with HIV (PLHIV) have a higher risk to be infected by TB as their immunocompromised status than that of HIV negative and as the cause of death in a quarter of PLHIV/AIDS4,5. Malnutrition and protein imbalance, i.e., in diabetes, can also impair the immune system and increase the risk of TB and TB-related death2,6. The daunting rise in cases of TB, HIV, and diabetes poses further major threats to public health worldwide. They were ranked as top diseases to cause high mortality in South East Asia (SEA), which accounted for deaths for 1.6 million, 940,000, and 30.3 million in 2017, respectively. The association between communicable and non-communicable diseases has been known for the past years, yet the optimization of the therapy remains scarce. Therefore, sustained and well-maintained healthcare approaches to make sure patients stay adherent and compliant to medication therapy are needed and remain of utmost importance.

Beyond the deadly combinations of the diseases and the improvement in disease treatments, an issue on the communication among the involved parties (e.g., physicians, pharmacists, and patients) needs to be marked crucial. Physicians and pharmacists have each specific role in the healthcare system, and the positive impacts of their collaboration have been established in several studies. The collaborative relationship between physicians and pharmacists accelerates the improvement of patient's therapy and thus provides a better quality of care. However, barriers in communications can still be noticed in the healthcare setting, especially in countries where the existence of pharmacists is limited. Time constraints and ineffective communication would be the significant points needing to be considered. This situation should be avoided as poor communication among them may lead to several negative impacts such as prescribing errors, treatment delay, unidentified adverse events, and even death7,8.

Over the last decades, mobile phone technology as a part of information and communication technology (ICT) has considerably been used in supporting diseases' treatments as a modality to improve medical care efficiency and adherence and to provide continuously updated clinical evidence. The ubiquity of mobile technologies, such as smartphones, enhances the ability to assess and improve general health. It has therefore created salient opportunities for the treatment and evaluation of a large number of common, intractable, expensive medical conditions. Such technologies in the healthcare setting can easily be accessed and are likely cost-effective, given its modest costs9. For example, a cost analysis of the use of mobile phones in Kenya revealed that text-message intervention in HIV treatment was cost-effective on the basic travel of expenses alone10. Conversely, concerns also have been expressed regarding the safety, confidentiality, quality of its content, and regulations on the use of mobile health applications11.

Much attention has been directed at the use of ICT in Indonesia due to the nations' unique geographic and socioeconomic characteristics. Indonesia is an archipelago country with 270 million population (population density of 140.08 individuals per square kilometer of land area)12. Being ranked 4th of countries with the highest population and the seventh largest country in terms of combined sea and land area worldwide, Indonesia is then believed to be one of the fastest growing markets for mobile phones in the SEA with 438.6 million mobile users. Having to mentioned the explanations above, the investigators, therefore, will research an easy-to-use - yet confidential and comprehensive - web-based healthcare application to be applied to high-risk patients; i.e., TB and HIV. By applying this web-based app to the specific population, the investigators hope to enhance the quality of care as well as the quality of life of such patients. The investigators will report on the findings and then discuss the future use of the web-based app.

With the complexity of drugs treatments in HIV and TB, treatment using mobile technologies is increasingly valued and becoming a trend over the past years. Technology that has a particular focus on patients' needs and ease-of-use and -access plays a significant role in the development of e-health and m-health. The proposed model of a secured mobile health application may promote patient's self-management and enhances adherence in chronic therapy exactly as it is easy-to-use, reducing patient's burden in accessing medication information and instructions, and providing the opportunity for direct communications with health providers in charge for each patient with access to mobile technologies. Consequently, medication errors and unnecessary paperwork in the healthcare system will be avoided as well as giving more time for healthcare providers to pay greater attention to delivering medical care effectively and efficiently.

The objective of the study is to conduct a usability testing of the web-based app in high-risk participants (HIV and TB patients). Usability testing will be conducted using a quantitative approach to evaluate the effectiveness, efficiency, and user satisfaction. After performing the usability testing of the web-based app on selected participants, investigators perform an in-depth interview to explore further problems, barriers, feedbacks, and potential advantages of the use of IeHS web-based app.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18 years old or more;
2. Acting as one of the following users: pulmonologist, internist, GP, pharmacists, and a patient who suffers from TB and/or HIV;
3. In case of a patient user: on drug treatment;
4. Use a smartphone and know how to use it;
5. Familiar with technology, particularly ICT;
6. Understand basic english;
7. Able to speak and communicate in Bahasa Indonesia;
8. Willing to participate and sign informed consent.

Exclusion Criteria:

1. A severe clinical condition that might impair the hearing or the seeing;
2. Unwillingness to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults males or females involved in HIV and TB treatment, i.e. physicians, pharmacists, HIV and/or TB patients.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Tasks completion success | during the simulation for each participant in 3 months of study period
  Effectiveness is defined by task completion success numbers of errors occur during the web-app simulation
Numbers of tasks errors | during the simulation for each participant in 3 months of study period
  Effectiveness is defined by task completion success numbers of errors occur during the web-app simulation
Average time to complete each task | during the simulation for each participant in 3 months of study period
  Efficiency is defined as level of efforts use by the study participant to complete the web-app simulation each task.
system usability scale (SUS) score | after half-an-hour of the web-app simulation during 3 months of study period
  IeHS satisfaction is defined through the SUS questionnaire which allows measurements of overall usability, allowing comparisons across a range of contexts and systems. SUS score is ranged from 0 (worst) to 100 (perfect).

SECONDARY OUTCOMES:
Participant experience using the IeHS web-based app | half an hour after web-based app simulation during 3 months of study period
  Participants/users are asked about their experiences and perceptions after the simulation regarding to the effectiveness, efficiency, satisfaction, obstacles, and IeHS potential use. These arguments will be collected qualitatively through in-depth interview.

CONTACTS AND LOCATIONS:
Overall Officials: Lusiana R Idrus, Master, Principal Investigator — Bekasi City Public Hospital
Locations (3):
- Indonesia (3):
  - Bekasi public hospital, Bekasi, West Java
  - Padang, Padang, West Sumatra
  - Jakarta, Jakarta

IPD SHARING:
Plan to Share IPD: Yes
Individual participants data are available for only 3 investigators (Lusiana, Najmatul Fitria, and Nahrul Hasan)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: November 2019 and will become available until publication
Access Criteria: Only for investigators

REFERENCES:
- [Background] GBD Tuberculosis Collaborators. The global burden of tuberculosis: results from the Global Burden of Disease Study 2015. Lancet Infect Dis. 2018 Mar;18(3):261-284. doi: 10.1016/S1473-3099(17)30703-X. Epub 2017 Dec 7. PMID 29223583
- [Background] Marais BJ, Lonnroth K, Lawn SD, Migliori GB, Mwaba P, Glaziou P, Bates M, Colagiuri R, Zijenah L, Swaminathan S, Memish ZA, Pletschette M, Hoelscher M, Abubakar I, Hasan R, Zafar A, Pantaleo G, Craig G, Kim P, Maeurer M, Schito M, Zumla A. Tuberculosis comorbidity with communicable and non-communicable diseases: integrating health services and control efforts. Lancet Infect Dis. 2013 May;13(5):436-48. doi: 10.1016/S1473-3099(13)70015-X. Epub 2013 Mar 24. PMID 23531392
- [Background] Glaziou P, Floyd K, Raviglione MC. Global Epidemiology of Tuberculosis. Semin Respir Crit Care Med. 2018 Jun;39(3):271-285. doi: 10.1055/s-0038-1651492. Epub 2018 Aug 2. PMID 30071543
- [Background] Podlekareva DN, Panteleev AM, Grint D, Post FA, Miro JM, Bruyand M, Furrer H, Obel N, Girardi E, Vasilenko A, Losso MH, Arenas-Pinto A, Cayla J, Rakhmanova A, Zeltina I, Werlinrud AM, Lundgren JD, Mocroft A, Kirk O; HIV/TB study group. Short- and long-term mortality and causes of death in HIV/tuberculosis patients in Europe. Eur Respir J. 2014 Jan;43(1):166-77. doi: 10.1183/09031936.00138712. Epub 2013 Jun 13. PMID 23766333
- [Background] WHO Treatment Guidelines for Drug-Resistant Tuberculosis, 2016 Update. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK390455/ PMID 27748093
- [Background] Workneh MH, Bjune GA, Yimer SA. Diabetes mellitus is associated with increased mortality during tuberculosis treatment: a prospective cohort study among tuberculosis patients in South-Eastern Amahra Region, Ethiopia. Infect Dis Poverty. 2016 Mar 21;5:22. doi: 10.1186/s40249-016-0115-z. PMID 27009088
- [Background] Free C, Phillips G, Watson L, Galli L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technologies to improve health care service delivery processes: a systematic review and meta-analysis. PLoS Med. 2013;10(1):e1001363. doi: 10.1371/journal.pmed.1001363. Epub 2013 Jan 15. PMID 23458994
- [Background] Patel AR, Kessler J, Braithwaite RS, Nucifora KA, Thirumurthy H, Zhou Q, Lester RT, Marra CA. Economic evaluation of mobile phone text message interventions to improve adherence to HIV therapy in Kenya. Medicine (Baltimore). 2017 Feb;96(7):e6078. doi: 10.1097/MD.0000000000006078. PMID 28207516